CLINICAL TRIAL: NCT00441779
Title: Retrospective Study of the Prevalence of Transfusion-Associated Microchimerism Following Traumatic Injury, Burns, and Elective Orthopedic Procedures
Brief Title: Transfusion-Associated Microchimerism in Previously Injured Individuals Who Received a Blood Transfusion
Status: Terminated | Type: Observational
Why Stopped: A separate study (similar subjects) identified transfusion-associated microchimerism only rarely, making this observational study impractical to conduct.
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 1378; 1R01HL083388 (NIH)
Record Dates: First submitted 2007-02-28; First posted 2007-03-01 (Estimated); Last update posted 2016-07-12 (Estimated); Status verified 2014-10

CONDITIONS: Chimerism; Blood Transfusion; Wounds and Injuries
Keywords: Microchimerism; Injuries; Burns; Orthopedic Surgery; Leukocytes
MeSH Terms: conditions — Wounds and Injuries; Burns

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Whole blood, plasma, peripheral blood mononuclear cells
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 1: Traumatic injury
- 2: Elective orthopedic surgery
- 3: Burn injury

SUMMARY:
Blood transfusions are frequently necessary in situations in which there is a large amount of blood loss. In some individuals who receive a blood transfusion, white blood cells from the donor's blood may remain in the body for years, a condition known as microchimerism. This study will evaluate the occurrence of microchimerism among the following three groups of individuals who previously received transfusions: 1) individuals with traumatic injuries; 2) individuals with burn injuries; and 3) individuals who underwent elective orthopedic operations.

DETAILED DESCRIPTION:
Approximately 10% to 15% of injured patients who receive blood transfusions experience a condition known as transfusion-associated microchimerism. This occurs when white blood cells, or leukocytes, from the donor's blood persist in the recipient long after the transfusion occurs. The genetically distinct donor cells can remain in the individual for decades, and may account for as many as 4% of the white blood cells in the recipient's body. This suggests that the donor cells are tolerated by the recipient's immune system. The purpose of this study is to compare the incidence of microchimerism among individuals with three different types of injuries: 1) traumatic injuries; 2) thermal, or burn, injuries; and 3) injuries resulting from elective orthopedic surgical procedures.

In this study, blood samples will be collected from individuals who were treated for traumatic injury, thermal injury, or elective orthopedic surgical procedures at the University of California at Davis Medical Center. Individuals who were treated from 2000 to 2003 and received a blood transfusion, as well as a control group of individuals who did not receive a transfusion, will be approached to enroll in the study. Individuals who agree to participate will have their blood analyzed for evidence of microchimerism. Information on health status, injury characteristics, hospital care, blood transfusion details, and blood donor characteristics will be collected from all participants.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized for traumatic injury, thermal injury, or an elective orthopedic surgical procedure from 2000 to 2003 at the University of California at Davis Medical Center
* Received at least 1 unit of transfused red blood cells

Exclusion Criteria:

* Currently incarcerated
* Inadequate decision-making capacity of the participant and no available surrogate decision-maker
* Prior bone marrow or solid organ transplantation
* Prior blood transfusion other than at the time of hospitalization
* Any history of an autoimmune disorder prior to hospitalization

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Previously hospitalized patients
Sampling Method: Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2008-08; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Microchimerism | 5-11 years after transfusion

CONTACTS AND LOCATIONS:
Overall Officials: Michael P. Busch, MD, PhD, Principal Investigator — Vitalant Research Institute
Locations (1):
- University of California, Davis, Medical Center, Sacramento, California, United States

REFERENCES:
- [Background] Utter GH, Owings JT, Lee TH, Paglieroni TG, Reed WF, Gosselin RC, Holland PV, Busch MP. Blood transfusion is associated with donor leukocyte microchimerism in trauma patients. J Trauma. 2004 Oct;57(4):702-7; discussion 707-8. doi: 10.1097/01.ta.0000140666.15972.37. PMID 15514522
- [Background] Utter GH, Owings JT, Lee TH, Paglieroni TG, Reed WF, Gosselin RC, Holland PV, Busch MP. Microchimerism in transfused trauma patients is associated with diminished donor-specific lymphocyte response. J Trauma. 2005 May;58(5):925-31; discussion 931-2. doi: 10.1097/01.ta.0000162142.72817.5c. PMID 15920405
- [Background] Lee TH, Paglieroni T, Utter GH, Chafets D, Gosselin RC, Reed W, Owings JT, Holland PV, Busch MP. High-level long-term white blood cell microchimerism after transfusion of leukoreduced blood components to patients resuscitated after severe traumatic injury. Transfusion. 2005 Aug;45(8):1280-90. doi: 10.1111/j.1537-2995.2005.00201.x. PMID 16078913